CLINICAL TRIAL: NCT07192783
Title: Effects of Lavender Oil Inhalation Applied to Patients With Primary Hypertension on Anxiety, Sleep Quality and Blood Pressure
Brief Title: The Effect of Lavender Inhalation on Anxiety, Sleep, and Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ardahan University (Other)
Responsible Party: Principal Investigator, Derya Şimşekli, Asist. Prof. Dr., Ardahan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ArdahanU-Şimsekli-DS-06
Record Dates: First submitted 2025-09-09; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Primary Hypertension
Keywords: primary hypertension; anxiety; sleep quality; blood pressure
MeSH Terms: conditions — Essential Hypertension; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: The study uses a parallel assignment design with two groups: an experimental group receiving lavender oil inhalation and a control group receiving routine care. Participants are randomly assigned to one of the two groups. The study is double-blinded: neither the participants, the researchers administering the intervention, nor the statisticians analyzing the data know group assignments. Outcomes (anxiety, sleep quality, and blood pressure) are measured before and after the one-month intervention period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, the interventionist, and the statistician are blinded. Patients are randomly assigned using simple randomization (odd-numbered to one group, even-numbered to the other). Group allocation (lavender oil or control) is determined by an independent nurse. Separate consent forms and coded data entry (groups as 1 and 2) ensure blinding is maintained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Participants receive lavender oil inhalation three times per week for one month (total of 12 sessions) in addition to routine care for primary hypertension. Anxiety, sleep quality, and blood pressure are assessed before and after the intervention.
  Interventions: Other: Lavender
- Routine care only (No Intervention): Participants in the control group continue their routine care and treatment for primary hypertension without receiving lavender oil inhalation. Anxiety, sleep quality, and blood pressure are assessed before and after the study period.

INTERVENTIONS:
Other: Lavender — Participants receive lavender oil inhalation three times per week for one month (total of 12 sessions) using a standardized diffuser. This intervention is provided in addition to routine care for primary hypertension. Outcomes measured include anxiety, sleep quality, and blood pressure before and after the intervention.
  Arms: experimental group

SUMMARY:
This study aims to determine the effects of lavender oil inhalation on anxiety, sleep quality, and blood pressure in patients with primary hypertension. The study is designed as a double-blind randomized controlled trial. The study population consists of patients presenting to the Cardiology Outpatient Clinic of Ardahan State Hospital. Participants are randomly assigned to an experimental group, which will receive a total of 12 lavender oil inhalations three times a week for one month, or to a control group, which will continue routine treatment and care. Data will be collected using the Hypertension Diagnostic Form, Beck Anxiety Inventory, and Pittsburgh Sleep Quality Index. Statistical analyses will be conducted to compare outcomes between the experimental and control groups.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of lavender oil inhalation on anxiety, sleep quality, and blood pressure in patients with primary hypertension. It is designed as a double-blind randomized controlled trial. Patients presenting to the Cardiology Outpatient Clinic of Ardahan State Hospital will be recruited for the study. Participants will be randomly assigned to an experimental group, which will receive 12 lavender oil inhalations three times a week for one month, or to a control group, which will continue routine care. Data will be collected using the Hypertension Diagnostic Form, Beck Anxiety Inventory, and Pittsburgh Sleep Quality Index. The study will assess whether lavender oil inhalation affects anxiety, sleep quality, and blood pressure in this population. Statistical analyses will be conducted to compare outcomes between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary hypertension
* Willing to participate in the study
* No allergy to lavender
* No olfactory impairments
* No history of psychiatric disorders

Exclusion Criteria:

* Communication difficulties
* Unwilling to participate
* Using other herbal or aromatherapy treatments
* History of sleep disorders affecting sleep quality (e.g., obstructive sleep apnea)
* Secondary hypertension or other chronic diseases
* Pregnant or breastfeeding
* Use of tobacco products

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-10-09 (Estimated); Study Completion 2025-10-09 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Baseline, Week 2, Week 4
  Measured using the Beck Anxiety Inventory (BAI) at baseline, week 2, and week 4. Higher scores indicate higher anxiety.
Blood Pressure | Baseline, Week 2, Week 4
  Measured using the Hypertension Diagnostic Form at baseline, week 2, and week 4. Includes systolic and diastolic measurements.

SECONDARY OUTCOMES:
Sleep quality | Baseline, Week 2, Week 4
  Measured using the Pittsburgh Sleep Quality Index (PSQI) at baseline, week 2, and week 4. Higher scores indicate poorer sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Ardahan State Hospital, Ardahan, Ardahan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality and privacy concerns of study participants.